CLINICAL TRIAL: NCT01961843
Title: Investigator-Initiated, Pilot Translational Study of Circulating Tumor Cells to Identify Predictive Factors of Response to Abiraterone Acetate in Men With Castration-Resistant Prostate Cancer
Brief Title: Abiraterone Acetate for Castrate Resistant Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard J. Lee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-209
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Castration Resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone acetate with Prednisone (Experimental): 1000 mg Abiraterone daily by mouth, 4 x 250 mg tablets Prednisone administered as 5 mg orally twice a day
  Interventions: Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone — Abiraterone acetate is an orally bioavailable inhibitor of steroid synthesis, specifically testosterone synthesis.
  Other Names: Abiraterone acetate; Zytiga
Drug: Prednisone — Prednisone is a synthetic corticosteroid that is co-administered with abiraterone acetate to offset the hypokalemia and hypertension side effects of abiraterone acetate.

SUMMARY:
This research study is a Pilot clinical trial. Pilot clinical trials often examine new tests (such as laboratory or radiology tests) in patients who receive either standard cancer treatments or new treatments that have been well-tested in many patients on other trials.

It is often difficult to determine how prostate cancer is going to behave when a new treatment is started. Physicians have no way to predict how a patient's tumor will respond to treatment. Although scientists have learned about changes that happen in tumors due to treatment, it is difficult to get cells from tumors because a biopsy (surgical procedure to remove a small piece of tissue) is needed.

This study will evaluate a method to detect tumor cells that are circulating in the blood without getting a biopsy. It is known that tumors shed a small number of cells into the blood stream every day. These are called circulating tumor cells or CTCs. Some early studies indicate the amount and type of CTCs in the blood can help determine the status of the tumor itself and the way it is responding to treatment. In this study, the investigators will examine protein levels in CTCs from patients' blood at different times before and after drug treatment to determine if they correlate with response to the drug. The new test will not affect whether subjects continue on the study drug.

Abiraterone acetate is a marketed drug that has been studied for the treatment of metastatic CRPC. It blocks the remaining or residual male hormones in the body that may be helping prostate cancer to grow. Abiraterone acetate is now FDA-approved for patients with metastatic CRPC who have not yet received docetaxel chemotherapy.

Abiraterone acetate has been used by a large number of participants in previous clinical trials. In most of these trials, participants with CRPC have been given abiraterone acetate with prednisone. Prednisone is a man-made hormone commonly referred to as a steroid. Prednisone has been approved in the US, Canada, and Europe for various disorders and diseases, such as asthma, Lupus and chronic obstructive lung disease. The combination of prednisone with abiraterone acetate has been approved for the treatment of CRPC. Prednisone together with abiraterone acetate will be given in this study in order to reduce or eliminate some side effects. Investigators will use patients' blood samples to study the genes (also called DNA) and their products (RNA and proteins) found in CTCs.

DETAILED DESCRIPTION:
If a patient agrees to participate in this research study, he will be asked to undergo some screening tests and procedures to confirm eligibility. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out the patient does not take part in the research study. These tests and procedures include: a medical history, physical exam, performance status, EKG, MUGA scan, bone scan, evaluation of the patient's disease, blood tests and a urine test. If these tests show that the patient is eligible to participate in the research study, he will begin the study treatment. If the patient does not meet the eligibility criteria, he will not be able to participate.

Once confirmed eligible to participate in the study, the patient will be started on the treatment. Patients will be seen in an outpatient setting. All patients will receive the study drugs, abiraterone acetate and prednisone. For the purposes of this description, study treatment will refer to abiraterone acetate in combination with prednisone.

Patients will take 4 tablets of abiraterone acetate by mouth daily. Patients will also take 1 tablet of prednisone by mouth twice a day. Patients will be given a study diary which includes instructions on how and when to take the study medication.

During the first two months in the study, patients will make about 3 visits to the clinic. Afterwards, patients will visit the clinic about once a month.

This study uses bone scans to assess worsening of subjects' prostate cancer (tumor progression) in the bones. Because arthritis can cause spots to appear on the bone scans, the scan is repeated a few weeks later. Cancer spots remain the same, but arthritis spots may disappear. Prostate Specific Antigen (PSA) tests can also be unreliable in the first few weeks after starting any new prostate cancer therapy. This is because the death of prostate cancer cells as a result of a new treatment can release PSA leading to an initial higher level in your blood. Such early rises in PSA can be mistaken for progression of a patient's cancer.

Cancer treatments can be divided into periods of time called cycles. A cycle in this study will last 28 days. At the start of each cycle of treatment, patients will be asked to visit the clinic to have regular pre-scheduled checkups and lab assessments. During Cycle 1 of this study, patients will be asked to come to the clinic twice for assessments, on Day 1 and Day 15. At these visits the study staff will talk to patients about the study in greater detail, perform all study visit procedures and provide the study treatment. The staff may also perform more tests and evaluations if needed.

If a subject continues to qualify for the study after Cycle 1, he will undergo a medical review, physical exam and blood sample on Day 1 of each cycle. Throughout the study, patients will be asked if you are experiencing any side effects. Subjects will be responsible for keeping your doctor informed if they feel they are having a reaction to the study treatment. In addition, subjects will be responsible for taking the medications on a daily basis as directed. It is very important to inform the treating clinician of any missed doses and the reasons why doses were missed, at each study visit. Patients will also be responsible for returning unused medication or the empty bottle at each study visit.

On Day 1 of Cycles 4, 7, 10 and every third cycle for as long as patients remain on study a blood sample for the CTC tests (about 2 tablespoons) will be collected. The following additional procedures will be done on Day 1 of Cycles 4, 7, 10 and every third cycle thereafter, and at Treatment Discontinuation: CT or MRI of abdomen and pelvis and bone scans.

After the final dose of study drug, patients will return for an End of Study Treatment Visit (15-28 days from treatment discontinuation). The tests completed at this end of study visit are the same as Cycle 1 Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Able to swallow the study drug whole as a tablet
* Willing to take abiraterone on an empty stomach
* Willing to use a method of birth control with adequate barrier protection
* Metastatic disease as documented by positive bone scan or metastatic lesions other than liver or visceral metastasis on CT, MRI
* Asymptomatic or mildly symptomatic from prostate cancer
* Surgically or medically castrated
* Previous anti-androgen therapy and progression after withdrawal
* Life expectancy of at least 6 months

Exclusion Criteria:

* Active infection or other medical condition that would make corticosteroid use contraindicated
* Uncontrolled hypertension
* Severe hepatic impairment
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic events in the past 6 months, severe or unstable angina, or NYHA Class III or IV heart disease
* Have any condition that, in the opinion of the investigator, would compromise the well being of the subject or the study or prevent the subject from meeting or performing study requirements
* Have poorly controlled diabetes
* Have a history of gastrointestinal disorders that may interfere with the absorption of the study agents
* Have a pre-existing condition that warrants long-term corticosteroid use in excess of study dose
* Have known allergies, hypersensitivity or intolerance to abiraterone acetate or prednisone or their excipients
* Pathologic finding consistent with small cell carcinoma of the prostate
* Liver, visceral organ or brain metastasis
* Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
* Radiation therapy for treatment of the primary tumor within 6 weeks of Cycle 1, Day 1
* Radiation or radionuclide therapy for treatment of metastatic CRPC tumor within 2 or 6 weeks, respectively, of Cycle 1, Day 1
* Previous treatment with ketoconazole for prostate cancer for greater than 7 days
* Prior systemic treatment with an azole drug
* Prior flutamide treatment within 4 weeks of Cycle 1, Day 1
* Bicalutamide, nilutamide within 6 weeks of Cycle 1, Day 1
* Active or symptomatic viral hepatitis or chronic liver disease
* History of a different malignancy except for the following circumstances: disease-free for at least 5 years and deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: basal cell or squamous cell carcinoma of the skin
* Administration of an investigational therapeutic within 30 days of Cycle 1, Day 1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-14; Primary Completion 2023-04-06 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of AR signaling in CTCs and correlation with response | 2 years
  To assess AR signaling in CTCs and correlate with PSA response and/or measurable disease response, if applicable. The investigators have developed a protein-based test to evaluate whether the AR signal is active ("AR-on") or inactive ("AR-off") or indeterminate ("AR-mixed"). The investigators will examine the AR signaling present in CTCs prior to and during abiraterone therapy. By correlating the baseline or post-treatment change in AR signaling with other measures of clinical benefit, the investigators aim to evaluate the use of AR signaling in CTCs to predict response to abiraterone. This may be applicable to other agents that target AR signaling.

SECONDARY OUTCOMES:
Change in number and proliferative fraction of CTCs with abiraterone treatment | 2 years
  The investigators will examine the number number and proliferative fraction of CTCs found in the blood of subjects prior to and during abiraterone treatment. Proliferation will be measured by Ki-67 staining. Baseline and post-treatment change in Ki-67 proliferative index will be correlated with other measure of clinical response to abiraterone.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No